CLINICAL TRIAL: NCT01227408
Title: Phase II Clinical Trial of Neoadjuvant Weekly Doxorubicin, Polyglutamate Paclitaxel, Capecitabine and Metronomic Chemotherapy in Breast Cancer
Brief Title: Neoadjuvant Doxorubicin, Polyglutamate Paclitaxel, Capecitabine and Metronomic Chemotherapy in Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrew due to funding issues
Sponsor: University of Southern California (Other)
Collaborators: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1B-08-7
Record Dates: First submitted 2009-01-08; First posted 2010-10-25 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: Patients with confirmed breast cancer for neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; paclitaxel poliglumex; Capecitabine; Cyclophosphamide; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Metronomic Chemotherapy (Experimental): Doxorubicin will be administered as an intravenous bolus, careful intravenous injection. PPX will be administerd as an intravenous 10 mins. infusion. Capecitabine and methotrexate will be taken orally twice a day. Cyclophosphamide will be taken orally once a day.
  Interventions: Drug: doxorubicin, paclitaxel poliglumex, capecitabine, cyclophosphamide, methotrexate

INTERVENTIONS:
Drug: doxorubicin, paclitaxel poliglumex, capecitabine, cyclophosphamide, methotrexate — doxorubicin 20mg/m2 weekly x 12 wks, cyclophosphamide 50 mg PO qd x 12 wks, methotrexate 2.5 mg PO bid d1,2 wkly x 12. One week later paclitaxel poliglumex 135mg/m2 IV every 3 wks plus capecitabine 825 mg/m2 PO bid x 14days x 4 cycles

SUMMARY:
The investigators propose to conduct a clinical trial of neoadjuvant treatment utilizing chemotherapy formulations with favorable toxicity profiles: weekly doxorubicin, PPX and capecitabine. It is expected this combination will at least maintain the efficacy of a traditional chemotherapy regimen but will be associated with less toxicity, particularly nausea, vomiting and alopecia. In order to accomplish this the investigators have designed a chemotherapy regimen whose components (or administration schedule) are associated with minimal or no alopecia and are also considered to have low emetogenic potential.

In an attempt to improve the efficacy of the regimen the investigators plan to study an alternate schedule of cyclophosphamide and methotrexate administration (metronomic chemotherapy) which appears to inhibit angiogenesis and therefore enhance the activity of conventional cytotoxic chemotherapy administered concurrently.

In this trial the investigators aim to determine the clinical and pathologic response rate of 12 weeks of doxorubicin followed by 4 cycles of PPX and capecitabine. Metronomic chemotherapy with cyclophosphamide and methotrexate will be administered during the 24 weeks of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* SWOG performance status of 0-2
* Projected life expectancy of at least 3 months
* Female age 18 years and over
* Provision of informed consent prior to any study-related procedures.
* Hormone receptor positive or negative tumor
* Her 2 neu negative tumor
* Negative pregnancy test for women of childbearing potential
* Patients must agree to use some form of contraception while on this study at initiation and for the duration of participation in the study. Sexually active males must also use a reliable and appropriate method of contraception. Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* ANC > 1500, Platelet count > 100,000, Hemoglobin > 9.0
* Serum creatinine < 1.5 mg/dl
* Hepatic function: Patients must have adequate liver functions: AST or ALT < 2.5 X upper limit of normal (ULN), alkaline phosphatase < 2.5 X upper limit of normal. Serum Bilirubin < 1.5 mg
* Peripheral neuropathy grade 0-1
* No other concomitant therapy directed at the cancer is allowed.

Exclusion Criteria:

* Serum bilirubin > 1.5 the upper limit of reference range (ULRR)
* Serum creatinine >1.5
* Prior therapy for this tumor.
* Clinical Congestive Heart Failure
* Women who are currently pregnant or breast feeding.
* Receipt of any investigational agents within 30 days prior to commencing study treatment
* Prior radiation must not have included ≥ 30% of major bone marrow containing areas (pelvis, lumbar spine)
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, lobular carcinoma in-situ of the breast (LCIS), or any other cancer from which the patient has been disease-free for 5 years. Patients with prior invasive breast cancer or ductal carcinoma in-situ (DCIS) are eligible if they have been disease free for 5 years and did not receive prior treatment with doxorubicin and/or a taxane.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02 (Estimated); Primary Completion 2010-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Response | At surgical resection on about week 30

SECONDARY OUTCOMES:
Toxicity | Every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States